CLINICAL TRIAL: NCT03028246
Title: A Feasibility Safety Study Using the ExAblate 4000 System in the Management of Benign Centrally-Located Intracranial Tumors Which Require Clinical Intervention in Pediatric and Young Adult Subjects
Brief Title: A Feasibility Safety Study of Benign Centrally-Located Intracranial Tumors in Pediatric and Young Adult Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT005
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Benign Centrally-Located Intracranial Tumors
Keywords: Hamartoma; Hypothalamic Hamartoma
MeSH Terms: conditions — Hamartoma; Hypothalamic hamartomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ExAblate 4000 System (Experimental): MR-Guided Focused Ultrasound
  Interventions: Device: ExAblate 4000 System

INTERVENTIONS:
Device: ExAblate 4000 System — Focused ultrasound
  Other Names: MRgFUS; HIFU; Focused Ultrasound; MR-Guided Focused Ultrasound; ExAblate Neuro System

SUMMARY:
The goal of this prospective, non-randomized, single-arm, feasibility study is to develop data to evaluate the safety and feasibility of ExAblate 4000 treatment of benign intracranial tumors which require clinical intervention in pediatric and young adult subjects.

Indication of Use: Ablation of benign intracranial tumors in children and young adults which are ExAblate accessible.

DETAILED DESCRIPTION:
The goal of this prospective, non-randomized, single-arm, feasibility study is to develop data to evaluate the safety and feasibility of ExAblate 4000 treatment of benign intracranial tumors which require clinical intervention in pediatric and young adult subjects.

Indication of Use: Ablation of benign intracranial tumors in children and young adults which are ExAblate accessible.

This is a feasibility study intended to collect data for use in the development of future studies. As such, no formal statistical hypothesis or hypothesis testing is proposed. The purpose of this study is to evaluate the safety and feasibility of managing benign brain tumor size using ExAblate 4000 treatment of progressing benign intracranial tumors which require clinical intervention in pediatric and young adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with benign (WHO grade I) centrally located intracranial tumors which require clinical intervention and are known to carry minimal hemorrhage risk
* Minimum head circumference will be 49cm
* Skull Density Ratio (SDR) should be ≥0.35
* Subjects should be on a stable dose of all condition-related medications for 30 days prior to study entry as determine by medical records
* Subjects and/or parent(s)/legal representative can provide accurate seizure diary log for the 30 days prior to FUS treatment and for the duration of the study

Exclusion Criteria:

* Subjects with unstable cardiac status that would increase anesthetic risk including
* Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV
* Subjects who are taking human growth hormone (hGH), also known as somatotropin
* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including vagus nerve stimulator, responsive neurostimulator, cardiac pacemakers, non-metallic shunts, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) or sedative medications
* Severely impaired renal function (estimated glomerular filtration rate <70% of normal GFR for age) or receiving dialysis
* Any history of clinically significant abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin, NSAIDs) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure; or, unable or unwilling to stop anticoagulant for the purpose of focused ultrasound procedure
* Use of valproate derivatives for seizure control within the preceding 2 weeks
* Known or suspected acute, active, or uncontrolled infection
* History of postnatal stroke or intracranial hemorrhage within 6 months
* Clinical suspicion of increased intracranial pressure (as evidenced by symptoms of obstruction: headache, nausea, vomiting, lethargy, and papilledema)
* Have participated in another interventional trial in the last 30 days
* History of immunocompromise, including subject who is HIV positive with incomplete viral suppression
* Known life-threatening systemic disease
* Subjects with suicidal ideation or previous suicide attempt within the past year
* Subjects with malignant brain tumors, or the presence of any ambiguous clinical features that could imply a malignant potential to the tumor, or for which a biopsy is necessary
* Subjects for whom histopathology is important for ongoing management
* Female subjects who are pregnant, breast feeding or planning to become pregnant during the study or are unwilling to practice birth control during participation in the study, if of child-bearing age

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events Safety and Tolerability | Post ExAblate Procedure through 12 Month Follow-up
  Safety will be assessed by tabulation of treatment related adverse events. All adverse events at least possibly procedure related will also be examined in detail for patterns of occurrence.
Measurement of Tumor Volume | Baseline through 12 Month Follow Up
  ExAblate procedure will demonstrate feasibility along with measurement of tumor volumes at follow-up as compared to the baseline MRI.

SECONDARY OUTCOMES:
Changes in the General Physical Exam | Baseline through 12 Month Follow Up
  Any changes in physical examination performed by a physician.
Changes in the Neurological Exam | Baseline through 12 Month Follow Up
  Any changes in neurological examination performed by the neurologist/neurosurgeon.
Confrontational Visual Field Testing | Baseline through 3 Month Follow Up
  Changes in confrontational visual field testing performed by a physician
Global Impression of Change-Clinician | Day 1 through 12 Month Follow Up
  Impression of change as the result of the treatment by a physician
Patient Global Impression of Change | Day 1 through 12 Month Follow Up
  Impression of change as the result of the treatment by the subject

OTHER OUTCOMES:
Change in Seizure Frequency | From baseline through 12 months after treatment
  The change in seizure frequency will be evaluated from baseline through 12 months after treatment.
QOLCE-55 | From baseline through 12 months after treatment
  The change in scores on the QOLCE-55 questionnaire will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: John Ragheb, MD, Principal Investigator — Miami Children's Research Institute - Nicklaus Children's Hospital
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: Undecided